CLINICAL TRIAL: NCT00794326
Title: Multicentric, Parallel, Controlled, Randomized, Single-blind Clinical Evaluation of New Low Sodium Peritoneal Dialysis Solution on Patients With Hypertension Treated With Continuous Ambulatory or Automated Peritoneal Dialysis
Brief Title: Clinical Evaluation of Low Sodium Peritoneal Dialysis (PD) Solution on Hypertensive Patients Treated With PD
Acronym: PDOne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1449; EudraCT 2007-005365-35
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Failure
Keywords: Chronic Kidney Failure; Peritoneal Dialysis; Low sodium solution; Hypertension; Total Body Water
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension | interventions — Dialysis Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDsol 12 (Experimental): Treatment with a peritoneal dialysis solution containing a low concentration of sodium.
  Interventions: Drug: Solution for Peritoneal Dialysis
- Gambrosol trio 40 (Active Comparator): Treatment with the peritoneal dialysis solution Gambrosol trio 40 isotonic bag (1.5%)
  Interventions: Drug: Solution for Peritoneal Dialysis

INTERVENTIONS:
Drug: Solution for Peritoneal Dialysis — Treatment with one bag per day during 6 months

SUMMARY:
The aim of this study is to assess the superiority of the new low sodium peritoneal dialysis (PD) solution PDsol 12 in comparison with a conventional, already marketed solution, Gambrosol trio 40, in the treatment of the hypertensive peritoneal dialysis patients with aim to decrease hypertension and to improve the sodium/water balance.

DETAILED DESCRIPTION:
Hypertension as well as sodium and water retention are common in end-stage renal disease patients on peritoneal dialysis and expose patients to left ventricular hypertrophy and increase cardiovascular mortality.

Moreover the poor control of dry weight and sodium/water balance results in increased morbidity. A previous low sodium study and computer simulations show that sodium removal can be improved with a low sodium fluid, which allows achieving a negative sodium balance without altering water balance.

The aim of this study is to assess whether treatment with one low sodium bag can substitute for one isotonic glucose bag every day in order to reduce the blood pressure and/or medication for hypertension, defined as the primary endpoint.

In order to evaluate the main criteria, blood pressure, a 24hours Ambulatory Blood Pressure Monitoring (ABPM) will be performed twice during the study, at Baseline and at 8 weeks of treatment, according to the EMEA guidance recommendations for anti-hypertensive treatments. In addition, the self measurement of blood pressure will be performed by patients at home during three consecutive days before each visit as well as in case of symptoms of hypotension.

The study is designed in three periods:

* Run-in period during 1 month: a reference product Gambrosol Trio 40, one bag/ day will be used by all patients. This period is dedicated to train the patient in using of study product, to stabilize the patient in the PD treatment and to randomize the patient, by performing the 24h ABPM.
* Efficacy & Safety period during 6 months: each patient will be treated with one of two product : PDsol 12 (studied product) or Gambrosol Trio 40 (reference product) during 6 months. The aim of this period is to evaluate the efficacy and long-term tolerance of new PD fluid.
* Follow-up period during 2 months: without treatment. This period is dedicated to ensure the safety of the patients after the study product treatment was stopped and to obtain the information about the reversibility of product effect.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure
* Stable patients on PD treatment
* Treatment at the study site for at least three months
* Treated in a CAPD program with a minimum of 3 bag exchanges with 6 or 7 days per week including at least one with duration of 4-6 hours, and at least one low strength bag per day, or in an APD program with at least one daytime exchange with duration of 4-6 hours using one low strength bag
* Hypertensive patients with high blood pressure at inclusion visit (Office SBP ≥ 140 and/or DBP ≥ 90 mmHg) or hypertensive patients receiving anti hypertensive medication including diuretics, disregarded blood pressure values
* Patients aged 18 years or more
* Written consent to participate in the study (informed consent)
* Able to use a three-compartment bag
* Life expectancy and expected technical survival ≥ 9 months

Exclusion Criteria:

* Low blood pressure (Office sitting SBP ≤ 120 mmHg and confirmed by ABPM < or = to 105 mean 24h SBP)
* Orthostatic hypotension defined as Systolic OBP with a drop of > 20mmHg and symptomatic after standing for at least 1 minute
* Natremia < 130 mmol/l, after two consecutive measurements
* Chronic arrhythmia
* Pregnancy or lactation
* Participation in other studies during the study period which may affect the outcome of the present study
* Peritonitis within one month prior to the study start
* Exit site and /or tunnel infection
* Patients unable to tolerate 2 L bag exchanges
* Patients on non-compatible PD system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary criterion is the ambulatory 24 h mean systolic blood pressure measurement and drug doses management after 2 months of treatment compared to Baseline. | At the beginning and after 8 weeks of treatment

SECONDARY OUTCOMES:
Measurement of Residual Renal Function | At the beginning, at two and six months of treatment
Follow-up of frequency of hyponatremia, of AE and SAE | During whole period of the study
Assessment of changes in sodium removal | At the beginning and at two months of treatment
Assessment of decrease in total body water (extra and intra cellular water)and of the body weigh changes | At the beginning, at two and at six months of treatment
Measurement of 24hours peritoneal clearance | At the beginning and at 2 months of treatment
Office systolic and diastolic blood pressure measurement at month 2 and 6 versus T0 | At the beginning, at two and six months of treatment
Office systolic and diastolic blood pressure measurement during follow up period | End of treatment, follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Simon Davies, Prof, Study Chair — University Hospital of North Staffordshire, Stoke-on-Trent, UK; Bengt Rippe, Prof, Study Chair — Lund University; Börje Haraldsson, Prof, Study Chair — Sahlgrenska University Hospital, Göteborg, Sweden; François Vrtovsnik, Prof, Study Chair — Bichat -Claude Bernard Hospital, Paris, France; Vedat Schwenger, Dr, Study Chair — Universitätsklinik University Hospital, Heidelberg, Germany
Locations (29):
- Rigshospitalet, Copenhagen, Denmark
- France (8):
  - CHU Saint-Jacques, Besançon
  - CHRU, Caen
  - Hospital of Chambéry, Chambéry
  - CH Colmar, Colmar
  - Calydial Dialysis Center, Irigny
  - Bichat-Claude Bernard Hospital, Paris
  - ARPDD, Reims
  - CHRU de Strasbourg, Strasbourg
- Germany (7):
  - KfH-Nierenzentrum, Cologne
  - KfH-Nierenzentrum am Krankenhaus Oststadt, Hanover
  - University Hospital of Heidelberg, Heidelberg
  - Nephrology center Offenburg, Offenburg
  - KfH-Nierenzentrum, Passau
  - PHV - Nephrologisches Zentrum Stuttgart, Stuttgart
  - KfH-Nierenzentrum Krankenhaus der Barmherzigen Brüder, Trier
- Sweden (7):
  - Södra Älvborgsläns Hospital, Borås
  - University Hospital of Sahlgrenska, Gothenburg
  - University Hospital of Lund, Lund
  - University Hospital of Malmö, Malmo
  - Skarborgs Hospital, Skövde
  - Karolinska University Hospital, Stockholm
  - Norra Älvsborgs Hospital, Trollhättan
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Southmead Hospital, Bristol
  - The Royal London Hospital, London
  - Royal Shrewsbury Hospital, Shrewsbury
  - University of North Staffordshire - Renal Medicine - Royal Infirmary, Stoke-on-Trent
  - Wolverhampton New Cross Hospital, Wolverhampton